Substitution Heuristic on Proportional Tasks NCT06762366 Version Date: 11/08/2024



Title of Research: Substitution in Adult Proportional Reasoning

Principal Investigator: Michelle Hurst, PhD

This online consent form is part of an informed consent process for research, and it will provide information that will help you decide whether you want to take part in the research. Ask questions if there is anything in the form that is not clear to you. If you decide to take part, instructions at the end of the document will tell you what to do next.

#### Who is conducting this research?

Michelle Hurst is the Principal Investigator of this research. A Principal Investigator has the overall responsibility for the conduct of the research. However, there are often other individuals who are part of the research team. Michelle Hurst may be reached at <a href="mailto:michelle.hurst@rutgers.edu">michelle.hurst@rutgers.edu</a> or (848) 445-1601 or via the anonymous messaging system within Prolific. This study is sponsored by the Eunice Kennedy Shriver National Institute of Child Health and Human Development, an institute of the National Institutes of Health.

#### Why is this research being done?

The purpose of the research is to understand how people think about different kinds of information, how the way we think changes across early childhood and into adulthood, and how external factors can change people's behavior and learning.

#### Who may take part in this research and who may not?

Adults between 18 and 64 years who are fluent in English may take part in this research.

# How long will the research take and how many participants will take part?

The expected length of this study is between 5 and 10 minutes. We expect to enroll a total of 300 participants across versions of this research project.

#### What will I be asked to do if I take part in this research?

You will be given information about quantities, visually (such as a set of items) or with symbols (such as a percentage) and asked to make judgements about the information. You might also be asked to answer survey questions about your preferences and personality and explain how you selected your choices for different parts of the study. Either before or during these activities, you may be given some instructions about what strategies you should use or be provided additional information related to the concepts in the activities.

#### What are the risks of harm or discomforts I might experience if I take part in this research?

There are no foreseen risks in participating in this study.

#### Are there any benefits to me if I choose to take part in this research?

There are no direct benefits to you.

#### What are my alternatives if I do not want to take part in this research?



Your alternative to participating in this research is to not take part in this research.

# Will there be any cost to me to take part in this study?

There are no costs to you for participating in this research.

# Will I be paid to take part in this study?

You will be paid at a rate of \$12 an hour, prorated for the expected advertised length of the study (for example, \$1.20 for a 6-minute study; \$1.60 for an 8-minute study). You will be paid via Prolific within 3 weeks of taking part with. We will not provide payment for incomplete studies, unless there was a technical error that was the fault of the researchers.

# How will information about me be kept private or confidential? What will happen to my information after the research is over?

The research is anonymous. No information will be collected that can identify who you are (e.g., your name, email address).

The non-identifiable data and information collected as part of this study may also be made publicly available on data repositories (e.g., the Open Science Framework at <a href="https://osf.io">https://osf.io</a>) and used by us or others in the future without obtaining additional permission from you. All data may be stored indefinitely (and for a minimum of 6-years) by the research team on secure cloud storage, password protected computers and hard drives, and in locked cabinets (in the case of physical or paper data).

Additionally, the research team may use or share your information collected or created for this study with the following people and institutions:

- The Rutgers University Institutional Review Board and Compliance Boards
- The Office for Human Research Protections in the U.S. Dept. of Health and Human Services
- National Institutes of Health

### **Certificate of Confidentiality**

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate does not stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate cannot be used to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate does not stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also does not prevent your information from being used for other research if allowed by federal regulations.

HRP-502a - Adult Consent for Interventional Research Template 10.30.23



Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about involvement in this research. It also does not prevent you from having access to your own information.

# What will happen if I do not wish to take part in the research or if I later decide not to stay in the research?

It is your choice whether to take part in the research. You may choose to take part, not to take part or you may change your mind and withdraw from the research at any time. If you do not want to enter the research or decide to stop taking part, your relationship with the research staff will not change, and you may do so without penalty and without loss of benefits to which you are otherwise entitled. Please note, however, that once you have submitted your responses, you may not be able to withdraw them as we will not know which ones are yours.

#### Who can I contact if I have questions?

If you have questions, concerns or complaints about the research, wish more information, you can contact the Principal Investigator, Dr. Michelle Hurst, and her research team at <a href="mailto:quadlab@psych.rutgers.edu">quadlab@psych.rutgers.edu</a>, or via the anonymous messaging system within Prolific.

If you have questions, concerns, problems, information or input about the research or would like to know your rights as a research subject, you can contact the Rutgers IRB or the Rutgers Human Subjects Protection Program via phone at (973) 972-3608 or (732) 235-2866 or (732) 235-9806 OR via email <a href="mailto:irboffice@research.rutgers.edu">irboffice@research.rutgers.edu</a>, or you can write us at 335 George Street, Liberty Plaza Suite 3200, New Brunswick, NJ 08901.

If you are 18 years of age or older, understand the statements above, and consent to take part in the study, click on the "I Agree" option and press the next button. If not, you may close this window or click the "I Do Not Agree" option and select next, which exit you from this screen/program.

| []I Agree |
|------------------------------------------------------------------------|
| [] I Do Not Agree |
| Please download or print a copy of this consent form for your records. |
| [NEXT BUTTON] |

Substitution Heuristic on Proportional Tasks NCT06762366 Version Date: 11/08/2024



Title of Research: Substitution in Adult Proportional Reasoning

Principal Investigator: Michelle Hurst, PhD

This online consent form is part of an informed consent process for research, and it will provide information that will help you decide whether you want to take part in the research. Ask questions if there is anything in the form that is not clear to you. If you decide to take part, instructions at the end of the document will tell you what to do next.

### Who is conducting this research?

Michelle Hurst is the Principal Investigator of this research. A Principal Investigator has the overall responsibility for the conduct of the research. However, there are often other individuals who are part of the research team. Michelle Hurst may be reached at <a href="mailto:michelle.hurst@rutgers.edu">michelle.hurst@rutgers.edu</a> or (848) 445-1601 or via the anonymous messaging system within Prolific. This study is sponsored by the Eunice Kennedy Shriver National Institute of Child Health and Human Development, an institute of the National Institutes of Health.

#### Why is this research being done?

The purpose of the research is to understand how people think about different kinds of information, how the way we think changes across early childhood and into adulthood, and how external factors can change people's behavior and learning.

#### Who may take part in this research and who may not?

Adults between 18 and 64 years who are fluent in English may take part in this research.

# How long will the research take and how many participants will take part?

The expected length of this study is between 5 and 10 minutes. We expect to enroll a total of 300 participants across versions of this research project.

#### What will I be asked to do if I take part in this research?

You will be given information about quantities, visually (such as a set of items) or with symbols (such as a percentage) and asked to make judgements about the information. You might also be asked to answer survey questions about your preferences and personality and explain how you selected your choices for different parts of the study. Either before or during these activities, you may be given some instructions about what strategies you should use or be provided additional information related to the concepts in the activities.

#### What are the risks of harm or discomforts I might experience if I take part in this research?

There are no foreseen risks in participating in this study.

#### Are there any benefits to me if I choose to take part in this research?

There are no direct benefits to you.

#### What are my alternatives if I do not want to take part in this research?



Your alternative to participating in this research is to not take part in this research.

# Will there be any cost to me to take part in this study?

There are no costs to you for participating in this research.

# Will I be paid to take part in this study?

You will be paid at a rate of \$12 an hour, prorated for the expected advertised length of the study (for example, \$1.20 for a 6-minute study; \$1.60 for an 8-minute study). You will be paid via Prolific within 3 weeks of taking part. We will not provide payment for incomplete studies, unless there was a technical error that was the fault of the researchers.

Bonus Payments: For part of the experiment, you may have the opportunity to receive bonus payments. You will receive more information about when these payments are available during the study.

# How will information about me be kept private or confidential? What will happen to my information after the research is over?

The research is anonymous. No information will be collected that can identify who you are (e.g., your name, email address).

The non-identifiable data and information collected as part of this study may also be made publicly available on data repositories (e.g., the Open Science Framework at <a href="https://osf.io">https://osf.io</a>) and used by us or others in the future without obtaining additional permission from you. All data may be stored indefinitely (and for a minimum of 6-years) by the research team on secure cloud storage, password protected computers and hard drives, and in locked cabinets (in the case of physical or paper data).

Additionally, the research team may use or share your information collected or created for this study with the following people and institutions:

- The Rutgers University Institutional Review Board and Compliance Boards
- The Office for Human Research Protections in the U.S. Dept. of Health and Human Services
- National Institutes of Health

#### **Certificate of Confidentiality**

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate does not stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate cannot be used to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate does not stop disclosures required by the federal Food and Drug Administration

HRP-502a - Adult Consent for Interventional Research Template 10.30.23



(FDA). The Certificate also does not prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about involvement in this research. It also does not prevent you from having access to your own information.

# What will happen if I do not wish to take part in the research or if I later decide not to stay in the research?

It is your choice whether to take part in the research. You may choose to take part, not to take part or you may change your mind and withdraw from the research at any time. If you do not want to enter the research or decide to stop taking part, your relationship with the research staff will not change, and you may do so without penalty and without loss of benefits to which you are otherwise entitled. Please note, however, that once you have submitted your responses, you may not be able to withdraw them as we will not know which ones are yours.

### Who can I contact if I have questions?

If you have questions, concerns or complaints about the research, wish more information, you can contact the Principal Investigator, Dr. Michelle Hurst, and her research team at <a href="mailto:quadlab@psych.rutgers.edu">quadlab@psych.rutgers.edu</a>, or via the anonymous messaging system within Prolific.

If you have questions, concerns, problems, information or input about the research or would like to know your rights as a research subject, you can contact the Rutgers IRB or the Rutgers Human Subjects Protection Program via phone at (973) 972-3608 or (732) 235-2866 or (732) 235-9806 OR via email <a href="mailto:irboffice@research.rutgers.edu">irboffice@research.rutgers.edu</a>, or you can write us at 335 George Street, Liberty Plaza Suite 3200, New Brunswick, NJ 08901.

If you are 18 years of age or older, understand the statements above, and consent to take part in the study, click on the "I Agree" option and press the next button. If not, you may close this window or click the "I Do Not Agree" option and select next, which exit you from this screen/program.

| [] I Agree |
|------------------------------------------------------------------------|
| [] I Do Not Agree |
| Please download or print a copy of this consent form for your records. |
| [NEXT BUTTON] |

HRP-502a - Adult Consent for Interventional Research Template 10.30.23